CLINICAL TRIAL: NCT04792931
Title: Adult Autoimmune Myopathies (MAIA): Clinical and Immunological Characterization, Constitution of a Patient Library
Brief Title: Adult Autoimmune Myopathies (MAIA)
Acronym: MAIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC20.0276
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Intervention Model Description: diagnosis and follow up of adult autoimmune myopathies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult Autoimmune Myopathies (Other): It is a description Autoimmune Myopathie cohort
  Interventions: Other: description of adult autoimmune myopathies

INTERVENTIONS:
Other: description of adult autoimmune myopathies — description of adult autoimmune myopathies

SUMMARY:
This study corresponds to a monocentric prospective cohort of adult patients presenting a suspicion of idiopathic inflammatory myopathy. It will allows the constitution of an organized collection of longitudinal clinical data as well as collection of biological samples, including blood sample, urine, stool and muscle specimen.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of Adult Inflammatory Myopathy
* Social security affiliation

Exclusion Criteria:

* Pregnant and lactating women
* Patients unable to consent
* Patients refusing to participate in the research.
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2030-05-20 (Estimated); Study Completion 2030-05-20 (Estimated)

PRIMARY OUTCOMES:
Distribution of lymphocytes subpopulations (B, T and TH-17) | 6 months
  Distribution of lymphocytes subpopulations (B, T and TH-17) according to the final diagnosis defined by a panel of experts

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de BREST, Brest, France